CLINICAL TRIAL: NCT07191132
Title: Integrating Multi-Modal Education to Improve Patient Compliance, Knowledge Retention, and Anxiety Reduction After Dental Extractions: A Randomized Controlled Trial
Brief Title: Multi-Modal Education to Improve Compliance, Knowledge Retention & Anxiety After Dental Extractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Malaysia (Other)
Responsible Party: Principal Investigator, Tan Su Keng, Associate Prof. Dr., Universiti Teknologi Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MDSC_UiTM
Record Dates: First submitted 2025-09-19; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Tooth Extraction; Postoperative Complications; Patient Compliance; Dental Anxiety; Patient Education as Topic
Keywords: Tooth Extraction; Postoperative Care; Patient Education; Dental Anxiety; Patient Compliance
MeSH Terms: conditions — Postoperative Complications; Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care providers performing the dental extractions were blinded to group allocation. Randomization occurred only after the extraction was completed, and the operating clinician was not involved in delivering post-operative instructions. Participants and the investigator providing instructions were not masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardised Verbal Instructions (Active Comparator): Participants receive the standardised verbal post-extraction care instructions delivered by a trained investigator using a calibrated script. No additional educational materials are provided.
  Interventions: Behavioral: Standardised Verbal Instructions
- Intervention - Verbal Instructions + PDEC-kit (Experimental): Participants receive the same standardised verbal post-extraction instructions as the control group, supplemented with the Post-Dental Extraction Care Kit (PDEC-kit). The kit includes:
  A 2-minute educational video
  Illustrated flashcards of dos and don'ts
  Live demonstration of gauze placement using a dental model
  Bilingual brochure (English and Bahasa Melayu), with QR code for digital access
  Interventions: Behavioral: Verbal Instructions + PDEC-kit

INTERVENTIONS:
Behavioral: Standardised Verbal Instructions — Participants receive verbal post-extraction care instructions delivered by a trained investigator using a calibrated script. The content includes guidance on bleeding control, diet, oral hygiene, activity restrictions, and medication use.
  Arms: Standardised Verbal Instructions
Behavioral: Verbal Instructions + PDEC-kit — Participants receive the same standardised verbal instructions as the control group, supplemented with the PDEC-kit. The kit includes a two-minute educational video, illustrated flashcards, a live gauze demonstration using a dental model, and a bilingual (English and Bahasa Melayu) illustrated brochure with QR code access to a digital version.
  Arms: Intervention - Verbal Instructions + PDEC-kit

SUMMARY:
The goal of this clinical trial is to learn whether using a new Post-Dental Extraction Care Kit (PDEC-kit) can help patients better understand and follow their post-extraction instructions, and whether it can also reduce dental anxiety, compared with verbal instructions alone. The study is being conducted among adult patients (18 years and older) undergoing routine tooth extractions under local anaesthesia at a university oral surgery clinic.

The main questions this study aims to answer are:

Does the PDEC-kit improve patients' knowledge retention about post-extraction care?

Does the PDEC-kit improve patient compliance with important post-extraction behaviours (e.g., medication use, diet, activity restrictions)?

Does the PDEC-kit reduce patient anxiety compared with standard verbal instructions?

Researchers will compare two groups of patients:

One group will receive the usual standardised verbal instructions.

The other group will receive the same verbal instructions plus the PDEC-kit.

Participants in the PDEC-kit group will:

Watch a short educational video on post-extraction care.

Review illustrated flashcards showing key "dos and don'ts."

Observe a live demonstration using a dental model to learn how to place and bite on gauze correctly.

Take home a bilingual brochure (English and Bahasa Melayu), also available via QR code.

All participants will be asked to answer short questionnaires about their knowledge, behaviour, and dental anxiety at three time points: before the extraction, immediately after receiving instructions, and one week later.

DETAILED DESCRIPTION:
Scientific Rationale

Tooth extraction is one of the most frequently performed dental procedures. Despite its routine nature, poor comprehension of post-operative instructions may lead to complications such as alveolar osteitis, infection, or delayed wound healing. Evidence from health communication research shows that patients retain only a small proportion of verbal-only instructions, particularly in settings of heightened anxiety. Multimedia learning theory (Mayer, 2021) suggests that simultaneous delivery of verbal, visual, and kinesthetic information enhances encoding and recall.

Building on this theory, the Post-Dental Extraction Care Kit (PDEC-kit) was developed. It integrates audiovisual, pictorial, and demonstration-based teaching into a structured package that supplements standard verbal guidance. The central hypothesis is that the PDEC-kit improves knowledge retention, compliance, and anxiety outcomes compared to verbal instructions alone.

Study Design Overview

This is a prospective, single-centre, two-arm, parallel-group randomized controlled trial. Participants are assigned to intervention or control groups in a 1:1 ratio. Allocation concealment was ensured using block randomisation with opaque, sequentially numbered envelopes. Operators performing extractions were blinded to allocation.

The sample size was determined by a priori power analysis using G*Power 3.1, based on a medium effect size (f = 0.25), α = 0.05, power = 0.80, and repeated measures across two groups. The minimum required sample was 86; recruitment was increased to 208 to account for attrition.

Intervention Details

Control arm: Standardised verbal post-extraction instructions delivered by a single calibrated investigator to minimise variability.

Intervention arm: Same standardised verbal instructions plus the PDEC-kit, which consists of:

Educational video (2 minutes): Demonstrates correct gauze placement, oral hygiene, and activity restrictions.

Illustrated flashcards: Show simplified dos and don'ts using pictorial reinforcement.

Live model demonstration: Gauze placement demonstrated on a dental model for kinesthetic learning.

Bilingual brochure (English and Bahasa Melayu): Provides at-home reference; a QR code enables access to a digital version.

All components were pilot-tested for clarity and developed by a multidisciplinary panel of oral surgeons, dental educators, and communication specialists.

Assessment Schedule

Data collection was performed at three points:

T0: Baseline (pre-extraction) - demographic data, knowledge baseline, and anxiety baseline.

T1: Immediately after instruction - post-intervention knowledge and anxiety assessments.

T2: One-week follow-up via telephone - reassessment of knowledge retention, anxiety, compliance, and complications.

Measurement Instruments

Knowledge retention: Four-item structured quiz (binary scoring).

Dental anxiety: Index of Dental Anxiety and Fear (IDAF-4C+, validated Malay version).

Compliance: Structured checklist covering analgesic use, diet, hygiene, activity, and smoking behaviour.

Pain: 10-point Likert scale.

Complications: Self-reported bleeding, infection, or alveolar osteitis, confirmed by clinic review where indicated.

Analytic Framework

Data were analysed using SPSS v29. Statistical procedures included:

Descriptive statistics for demographic and baseline variables.

Independent-samples t-test for between-group comparisons.

Paired-samples t-test for within-group pre-post changes.

Repeated measures ANOVA (Greenhouse-Geisser correction applied when sphericity violated).

Chi-square test for categorical variables (compliance, complication rates).

Spearman's correlation for anxiety-pain association. Significance threshold: p < 0.05.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older
* Scheduled for routine, non-surgical extraction of one or two adjacent permanent teeth
* Able to read and understand either English or Bahasa Melayu

  -=Classified as American Society of Anesthesiologists (ASA) physical status I or II
* Provide written informed consent

Exclusion Criteria

* Previous participation in this study
* ASA physical status III or higher
* History of diagnosed anxiety disorders, depression, or learning disabilities
* Requirement for surgical, complex, or multiple extractions
* Procedures expected to be difficult or requiring assistance from a supervising specialist
* Inability to understand or follow study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Knowledge Retention of Post-Extraction Care | Baseline (pre-extraction, T0), immediately after instruction (T1), and one-week post-operatively (T2).
  Knowledge assessed using a structured four-item post-extraction care quiz (binary scoring, correct/incorrect). Higher scores indicate better knowledge retention.

SECONDARY OUTCOMES:
Dental Anxiety (IDAF-4C+) | Baseline (T0), immediately after instruction (T1), and one-week post-operatively (T2).
  Level of dental anxiety measured using the validated Index of Dental Anxiety and Fear (IDAF-4C+), including core, phobia, and stimulus modules.
  Structure:
  * Core module (8 items): Each item is scored on a 5-point Likert scale (1 = Disagree to 5 = Strongly agree).
  * Phobia module (5 items, Yes/No): Screens for dental phobia.
  * Stimulus module (10 items): Rates fear related to specific dental stimuli and situations on a 5-point scale (1 = Not at all to 5 = Very much).
  Scoring:
  Core module total score range: 8 (minimum) to 40 (maximum). Interpretation: Higher scores indicate a worse outcome (greater dental anxiety/fear).
  Phobia and stimulus modules are analyzed separately; higher values indicate greater anxiety/fear or avoidance.
Patient Compliance with Post-Operative Instructions | One-week post-operatively (T2).
  Adherence to specific behaviours (analgesic use, diet, oral hygiene, activity restriction, and smoking cessation) assessed using a structured compliance checklist adapted from Shenoi et al. (2021).

OTHER OUTCOMES:
Self-Reported Pain | Baseline (T0), immediately after instruction (T1), and one-week post-operatively (T2).
  Pain severity assessed using a 10-point Likert numerical rating scale (0 = no pain; 10 = worst possible pain).
Post-Operative Complications | One-week post-operatively (T2).
  Self-reported complications including bleeding, infection, or alveolar osteitis, confirmed by clinic follow-up where necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mohammad, BDS, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- Faculty of Dentistry Universiti Teknologi MARA, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in published articles will be made available to other researchers.
  De-identified individual participant data underlying the primary and secondary outcomes reported in the main publication.
  How to access data: Requests should be submitted to the corresponding author (Tan Su Keng, Centre of Studies for Oral & Maxillofacial Surgery, Universiti Teknologi MARA). Approved requests will require a signed data use agreement, and data will be shared via secure e
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of the primary study results and for up to 5 years thereafter.
Access Criteria: Data will be available to researchers with a methodologically sound proposal, subject to approval by the principal investigator and UiTM Research Ethics Committee.

REFERENCES:
- [Background] Klueber KM, Langdon HL, Barnwell Y. The morphology of the vertical and transverse intrinsic musculature of the tongue in the 15-week human fetus. Acta Morphol Neerl Scand. 1979 Dec;17(4):301-10. PMID 539473
- [Background] Mayer, R. E. (2021). The Cambridge Handbook of Multimedia Learning (2nd ed.). Cambridge University Press. https://doi.org/10.1017/CBO9781139547369
- [Background] Svensson L, Hakeberg M, Wide U. Evaluating the validity of the Index of Dental Anxiety and Fear (IDAF-4C+) in adults with severe dental anxiety. Eur J Oral Sci. 2020 Oct;128(5):423-428. doi: 10.1111/eos.12731. Epub 2020 Aug 16. PMID 33463781
- [Background] Fathima T, Kumar MPS. Evaluation of quality of life following dental extraction. J Adv Pharm Technol Res. 2022 Nov;13(Suppl 1):S102-S107. doi: 10.4103/japtr.japtr_361_22. Epub 2022 Nov 30. PMID 36643114
- [Background] Dignam P, Elshafey M, Jeganathan A, Foo M, Park JS, Ratnaweera M. Prevalence and Factors Influencing Post-Operative Complications following Tooth Extraction: A Narrative Review. Int J Dent. 2024 May 9;2024:7712829. doi: 10.1155/2024/7712829. eCollection 2024. PMID 38756385
- [Background] Alvira-Gonzalez J, Gay-Escoda C. Compliance of postoperative instructions following the surgical extraction of impacted lower third molars: a randomized clinical trial. Med Oral Patol Oral Cir Bucal. 2015 Mar 1;20(2):e224-30. doi: 10.4317/medoral.20121. PMID 25475774
- [Background] Udeabor SE, Heselich A, Al-Maawi S, Alqahtani AF, Sader R, Ghanaati S. Current Knowledge on the Healing of the Extraction Socket: A Narrative Review. Bioengineering (Basel). 2023 Sep 29;10(10):1145. doi: 10.3390/bioengineering10101145. PMID 37892875
- [Background] Shenoi RS, Rajguru JG, Parate SR, Ingole PD, Khandaitkar SR, Karmarkar JS. Compliance of postoperative instructions following the surgical extraction of impacted lower third molars. Indian J Dent Res. 2021 Jan-Feb;32(1):87-91. doi: 10.4103/ijdr.IJDR_323_20. PMID 34269243
- [Background] Ploghaus A, Narain C, Beckmann CF, Clare S, Bantick S, Wise R, Matthews PM, Rawlins JN, Tracey I. Exacerbation of pain by anxiety is associated with activity in a hippocampal network. J Neurosci. 2001 Dec 15;21(24):9896-903. doi: 10.1523/JNEUROSCI.21-24-09896.2001. PMID 11739597
- [Background] Ikmalhisam, N., Aziz, N., Mah, M., Jamaluddin, T., Wahab, H., Mohammad, M., & Tan, S. (2021). Delivery of Post-Dental Extraction Care Instructions with the Aid of a Novel Educational Kit: The UiTM Dental Students' Perspective. ESTEEM Academic Journal, 17, 135-146.
- [Background] Houts PS, Witmer JT, Egeth HE, Loscalzo MJ, Zabora JR. Using pictographs to enhance recall of spoken medical instructions II. Patient Educ Couns. 2001 Jun;43(3):231-42. doi: 10.1016/s0738-3991(00)00171-3. PMID 11384821
- [Background] Dingley C, Daugherty K, Derieg MK, Persing R. Improving Patient Safety Through Provider Communication Strategy Enhancements. In: Henriksen K, Battles JB, Keyes MA, Grady ML, editors. Advances in Patient Safety: New Directions and Alternative Approaches (Vol. 3: Performance and Tools). Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK43663/ PMID 21249923
- [Background] Choi SH, Won JH, Cha JY, Hwang CJ. Effect of Audiovisual Treatment Information on Relieving Anxiety in Patients Undergoing Impacted Mandibular Third Molar Removal. J Oral Maxillofac Surg. 2015 Nov;73(11):2087-92. doi: 10.1016/j.joms.2015.06.175. Epub 2015 Jul 8. PMID 26212090
- [Background] Baharuddin IH, Arifin WN, Kueh YC, Rahman NA. Adaptation and Validation of the Malay Version of the Index of Dental Anxiety and Fear (IDAF-4C+) for Malaysian Secondary School Children. Malays J Med Sci. 2018 May;25(3):111-119. doi: 10.21315/mjms2018.25.3.11. Epub 2018 Jun 28. PMID 30899192
- [Background] Armfield JM. Development and psychometric evaluation of the Index of Dental Anxiety and Fear (IDAF-4C+). Psychol Assess. 2010 Jun;22(2):279-87. doi: 10.1037/a0018678. PMID 20528055